CLINICAL TRIAL: NCT02006264
Title: Phase 1 Safety and Pharmacokinetic Study of Polyurethane Tenofovir Disoproxil Fumarate Vaginal Ring
Brief Title: Safety and Pharmacokinetics (PK) of a Polyurethane Tenofovir Disoproxil Fumarate (TDF) Vaginal Ring
Acronym: TDF IVR-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Marla Keller, Prof. Dept of Medicine, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2013-329; U19AI076980 (NIH)
Record Dates: First submitted 2013-11-19; First posted 2013-12-10 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: HIV

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- TDF Intravaginal Ring (Active Comparator): Tenofovir Disoproxil Fumarate intravaginal ring (TDF-IVR) is a white (with clear segment), flexible torus-shaped device with an inner core compartment comprised of TDF (86 wt% of formulation) and Sodium Chloride (NaCl) (14 wt% of formulation). The intravaginal ring will be worn continuously for 14 days. It will be inserted into the vagina following cessation of participant's menses at Visit 3 and removed at Visit 7.
  Interventions: Drug: TDF Intravaginal Ring
- Placebo Intravaginal Ring (Placebo Comparator): The placebo intravaginal ring (IVR) is a clear, flexible torus-shaped device with an inner core which contains sodium chloride (NaCl). The intravaginal ring will be worn continuously for 14 days. It will be inserted into the vagina following cessation of participant's menses at Visit 3 and removed at Visit 7.
  Interventions: Drug: Placebo Intravaginal Ring

INTERVENTIONS:
Drug: TDF Intravaginal Ring — The TDF IVR intravaginal ring is formulated using flexible outer tubing, comprised of hydrophilic, aliphatic polyether urethane, and an inner core compartment comprised of 86% w/w TDF and 14% w/w sodium chloride (NaCl). The TDF intravaginal ring will be worn continuously for 14 days. It will be inserted into the vagina following cessation of participant's menses at Visit 3 and removed at Visit 7.
  Other Names: TDF IVR
  Arms: TDF Intravaginal Ring
Drug: Placebo Intravaginal Ring — The placebo ring is formulated using flexible outer tubing, comprised of hydrophilic, aliphatic polyether urethane, and an inner core comprised of sodium chloride (NaCl). The Placebo intravaginal ring will be worn continuously for 14 days. It will be inserted into the vagina following cessation of participant's menses at Visit 3 and removed at Visit 7.
  Other Names: Placebo
  Arms: Placebo Intravaginal Ring

SUMMARY:
This prospective, randomized, single-blinded, placebo controlled trial will examine the safety and pharmacokinetics (PK) of a polyurethane tenofovir disoproxil fumarate (TDF) vaginal ring when used continuously for 14 consecutive days.

The primary objective is to assess the safety of TDF vaginal rings when used continuously for 14 days by healthy, HIV-uninfected, sexually abstinent women, as compared with a placebo vaginal ring.

DETAILED DESCRIPTION:
Tenofovir disoproxil fumarate (TDF) is a prodrug of TFV (tenofovir), an adenosine nucleoside monophosphonate (nucleotide) derivative with potent antiretroviral (ARV) activity. TDF permeates cells more rapidly than TFV resulting in increased intracellular accumulation of TFV-diphosphate (TFV-DP), the active metabolite. TDF is more potent than TFV and inhibits HIV-1 (Human Immunodeficiency Virus-1)and herpes simplex virus type 2 (HSV-2) infection in cell and tissue culture models at approximately 100-fold lower concentrations than TFV, suggesting that it may be an excellent candidate for prevention of HIV. TDF is licensed for the treatment of HIV-1 infection in the US, the European Union, Middle East, and Africa.

The study will take place at the Albert Einstein College of Medicine in Bronx, New York, USA. Each participant will receive an IVR (intravaginal ring) containing TDF or a placebo ring. The vaginal ring will be worn continuously for 14 days. It will be inserted into the vagina following cessation of participant's menses, by the study clinician at Visit 3 and removed by the study clinician at Visit 7. Each participant will be followed for 7 days following ring removal.

It is hypothesized that both the TDF IVR and placebo IVR will be safe and well tolerated among healthy, sexually abstinent women on combined-hormonal contraception. The null hypothesis is that there will be no difference in the safety profile between the active product and the placebo.

Careful assessments of safety, including systemic and genital tract, will be undertaken with special consideration for issues related to irritation and systemic toxicity. The design of the study will allow safety comparisons of TDF ring to a placebo ring. A 14-day safety and PK study is proposed for this first-in-human study per FDA (For and Drug Administration) guidance. The study duration was carefully selected to control risk to the study participants. TFV 1% vaginal gel has been extensively tested in clinical trials at higher doses (8-fold dose margin) than the predicted dose delivered by the TDF IVR-001 study, and the TFV gel showed no significant adverse events at this higher dose in thousands of women.

Given the drug release kinetics observed in vitro and in NHP (non-human primate) studies, TDF and TFV (formed following hydrolysis of the prodrug TDF) concentrations in cervicovaginal fluid (CVF) are expected to reach steady state within a few days and maintain steady state concentrations for the duration of the planned 14 days of ring use. Sampling at multiple time points and sites (vaginal, cervical, rectal and blood) will provide information on drug distribution, kinetics, and, by sampling after ring removal on Day 14, how long drug persists. The latter may be important as behavior studies suggest that some women may remove a ring at time of menses or around sex. To capture systemic absorption, blood will be sampled to determine drug concentrations in blood plasma and PBMCs (peripheral blood mononuclear cells). To capture the concentrations of drug within the genital tract, CVF will be sampled using Dacron swabs of the introitus, ectocervix, and area adjacent to the ring. Rectal sampling with swabs will also be obtained if participants consent to the procedure to determine drug concentrations in the rectum. Sampling at different sites (proximal and distal to the ring) will provide important information as to how well drug permeates throughout the genital tract. Cervical tissue sampling will be highly informative given that it is the likely site of drug action. However, biopsies must be taken sparingly for several reasons: they are uncomfortable to some and alter the healing process. Accordingly, two baseline biopsies will be taken prior to randomization and ring insertion to confirm absence of study drug and for PD studies. Subsequent biopsies for PK (pharmacokinetics) and PD (pharmacodynamics) studies will be delayed until the ring is removed. Following TDF IVR removal a third biopsy will be obtained for PK studies. Two cervical biopsies will be obtained following placebo IVR removal for PD studies and to blind safety data. The study will not be double-blinded because the TDF and placebo rings are not identical in appearance. Therefore, the study clinician will be able to collect two biopsies from participants in the placebo group and three biopsies from participants in the TDF ring group after ring removal. In order to maintain participant blinding, all participants will be informed that two biopsies will be taken before ring insertion and 2-3 biopsies will be taken after ring removal. Paired biopsies will provide the best data, as it will avoid inter-individual variability; both sets of cervical biopsies (pre- and post-IVR use) will be obtained during the second half of the participant's menstrual cycle (cycle days 18-23), which is prior to menses. Cervical biopsies will be obtained without local anesthetic. Participants may take acetaminophen before and/or after the biopsies are collected if desired.

Primary Objective:

• Assess the safety of TDF IVR when used continuously for 14 days by healthy, HIV-uninfected, sexually abstinent women, as compared with the placebo IVR

Secondary Objective:

• Examine systemic and genital tract PK of TDF release during and after 14 days of continuous use of a reservoir-type IVR containing TDF

Exploratory Objectives:

* Evaluate the acceptability of and adherence to the study IVR
* Evaluate the PD during and after 14 days of continuous use of a reservoir-type IVR containing TDF by measuring the antiviral activity of genital tract secretions ex vivo and challenging biopsy tissue with virus
* Examine the impact of the study IVR on genital tract mucosal immunity and the vaginal microbiota
* Examine the PK of TDF and TFV in rectal fluid during and after 14 days of continuous use of a reservoir-type TDF IVR
* Evaluate mechanical properties and drug content following 14 days of continuous use of reservoir-type IVRs

This is a single-site, two-arm, randomized single-blind, placebo-controlled trial. The study population will include approximately 30 healthy, 18-45 year old women who are HIV-uninfected, non-pregnant, sexually abstinent and using adequate contraception, as described in the protocol. This sample size was chosen with the goal of having 12 women per group complete the study and includes additional women to account for participants who may not complete the study or are lost to follow-up. Only female volunteers will be recruited since an IVR can only be used by women and the endpoints require genital sampling. To ensure participants are protected from pregnancy during study participation, to minimize variability among contraceptive methods, and to ensure adequate time between menses for ring use and sample collection, all volunteers must be using low-dose combined hormonal contraceptive pills. As this is a first-in-human trial of an intravaginal TDF ring, only healthy women will be recruited and will be asked to wear a TDF or placebo IVR for 14 days.

The approximate time to complete study enrollment is expected to be 9 months. Two study groups are planned. Both groups will be assigned to complete a total of 9 study visits: (Screening [Visit 1], Enrollment [Visit 2], Days 0 [Visit 3], 1 [Visit 4], 3-5 [Visit 5], 7 [Visit 6], 14 [Visit 7], 16-18 [Visit 8], 21 [visit 9]). A Safety Call will also be conducted on Day 10 of the study.

The two study groups are:

1. Reservoir-type TDF IVR group;
2. Reservoir-type polyurethane IVR group;

The expected duration for participants is approximately 5 - 10 weeks (including a screening visit, an enrollment visit, two weeks of continuous IVR use, and one week following IVR removal). Participants will undergo Visit 2 within 45 days of screening. No study data will be collected after the Final Study/Early Termination Visit unless the participant is pregnant at the Final Study/Early Termination Visit. Participants who have AEs (adverse events) at the Final Study/Early Termination Visit that have not resolved or stabilized will be followed beyond the Final Study/Early Termination Visit until a clinically acceptable resolution of the AE(s) is confirmed and documented. Clinical acceptability of resolution will be determined by the PL (Program Leader) in consultation with the Protocol Safety Review Team (PSRT). Participants who are pregnant at the Final Study/Early Termination Visit may be followed in accordance with procedures described in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* General good health (by volunteer history and per investigator discretion) without any clinically significant systemic disease (including, but not limited to significant liver disease/hepatitis, gastrointestinal disease, kidney disease, thyroid disease, osteoporosis or bone disease, and diabetes)
* Willing to give voluntary consent, sign an informed consent form and comply with study procedures as required by the protocol
* HIV-uninfected based on testing performed by study staff during screening procedures
* Using low dose combined (estrogen and progesterone-containing) oral contraceptive pills (does not include extended-cycle, 24 and 28-day active pill regimens). Per participant report must be using this contraceptive method with no change in the prior 3 months and intending to use same method for the duration of study participation.
* Currently have a regular 28-day menstrual cycle on combined oral contraceptive pills.
* Normal Pap test at screening or appropriately documented history of Pap test and completed follow-up of any abnormal pap tests consistent with American Congress of Obstetricians and Gynecologists (ACOG) practice guidelines #99 and #109.
* Agrees not to participate in other research studies involving drugs, medical devices, or vaginal products for the duration of study participation.
* Able and willing to refrain from inserting any non-study vaginal products or objects into the vagina for the 48 hours prior to Visit 2 throughout the duration of the study.
* Able and willing to abstain from oral, vaginal and anal sex for 48 hours prior to Visit 2 throughout the duration of the study.

Exclusion Criteria:

Women must meet none of the following criteria prior to genital sampling at Visit 2:

* Known adverse reaction to polyurethane or to any components of the study product or allergy to both silver nitrate and Monsel's solution.
* Hepatitis B infection (defined as positive hepatitis B surface antigen).
* Chronic, recurrent, and/or acute vulvar or vaginal symptoms (pain, irritation, spotting, etc.).
* Known bleeding disorder that could lead to prolonged or continuous bleeding with biopsy.
* Pregnant or intending to become pregnant during the period of study participation.
* Currently breastfeeding or having breastfed an infant in the last two months, or planning to breastfeed during the course of the study.
* Menopause.
* History of unexplained or unresolved intermenstrual bleeding in the 3 months prior to screening.
* History of gynecological procedures (including genital piercing) on the external genitalia, vagina or cervix in the last 14 days.
* Hysterectomy.
* Use and/or anticipated use during the study period of an intravaginal or intrauterine device.
* Systemic use in the last 2 weeks or anticipated use during the study period of any of the following: corticosteroids, antibiotics, antifungals, antivirals, anticoagulants or antiretrovirals.
* Grade 1 or higher laboratory abnormality, per the August 2009 update of the Division of AIDS, National Institute of Allergy and Infectious Disease (DAIDS) Table for Grading the Severity of Adverse Events (AEs).
* In the last six months, diagnosed with or treated for any sexually transmitted infection (STI).
* Reproductive tract infection (RTI) or pelvic inflammatory disease (PID) requiring treatment per current CDC (Center for Disease Control and Prevention) guidelines at Screening or Enrollment.
* Positive test for Trichomonas vaginalis, Neisseria gonorrhea or Chlamydia trachomatis at screening.
* Reactive test for syphilis at screening.
* At Screening or Enrollment, has a clinically apparent Grade 1 or higher pelvic exam finding (observed by study clinician or designee) per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Addendum 1, Female Genital Grading Table for Use in Microbicide Studies.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11-19; Primary Completion 2014-11-06 (Actual); Study Completion 2014-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marla J Keller, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

REFERENCES:
- [Background] Smith JM, Rastogi R, Teller RS, Srinivasan P, Mesquita PM, Nagaraja U, McNicholl JM, Hendry RM, Dinh CT, Martin A, Herold BC, Kiser PF. Intravaginal ring eluting tenofovir disoproxil fumarate completely protects macaques from multiple vaginal simian-HIV challenges. Proc Natl Acad Sci U S A. 2013 Oct 1;110(40):16145-50. doi: 10.1073/pnas.1311355110. Epub 2013 Sep 16. PMID 24043812
- [Background] Mesquita PM, Rastogi R, Segarra TJ, Teller RS, Torres NM, Huber AM, Kiser PF, Herold BC. Intravaginal ring delivery of tenofovir disoproxil fumarate for prevention of HIV and herpes simplex virus infection. J Antimicrob Chemother. 2012 Jul;67(7):1730-8. doi: 10.1093/jac/dks097. Epub 2012 Mar 30. PMID 22467632

RESULTS

PARTICIPANT FLOW:
Groups:
- TDF Intravaginal Ring: TDF Intravaginal Ring (TDF-IVR)
  The TDF (tenofovir disoproxil fumarate) IVR (intravaginal ring) has an inner core compartment comprised of 86% w/w (weight by weight) TDF and 14% w/w sodium chloride (NaCl). The TDF intravaginal ring will be worn continuously for 14 days. It will be inserted into the vagina following cessation of participant's menses at Visit 3 and removed at Visit 7.
- Placebo Intravaginal Ring: Placebo Intravaginal Ring (Placebo IVR)
  The placebo intravaginal ring (IVR) has an inner core which contains sodium chloride (NaCl). The intravaginal ring will be worn continuously for 14 days. It will be inserted into the vagina following cessation of participant's menses at Visit 3 and removed at Visit 7.
Period: Overall Study
Arm/Group | TDF Intravaginal Ring | Placebo Intravaginal Ring
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- TDF Intravaginal Ring: TDF Intravaginal Ring (TDF IVR)
- Placebo Intravaginal Ring: Placebo Intravaginal Ring (Placebo IVR)
- Total: Total of all reporting groups
Arm/Group | TDF Intravaginal Ring | Placebo Intravaginal Ring | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (7.1) | 28.2 (5.7) | 29.65 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Grade 1 Genitourinary Events or Higher as Defined by the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events
Description: Grade 1 or higher Genitourinary events as defined by the DAIDS (Division of AIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events during the trial period judged to be related to study product
Time Frame: 14 days of vaginal ring use
Measure: Number; unit: Adverse events
Arm/Group | TDF Intravaginal Ring | Placebo Intravaginal Ring
Number analyzed (Participants) | 15 | 15
Adverse events | 7 | 1

2. Primary Outcome: Grade 2 or Higher Adverse Events as Defined by the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events
Description: Grade 2 or higher systemic and local Adverse Events as defined by the Division of Aids (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events during the trial period
Time Frame: 14 days of vaginal ring use
Measure: Number; unit: Adverse events
Arm/Group | TDF Intravaginal Ring | Placebo Intravaginal Ring
Number analyzed (Participants) | 15 | 15
Adverse events | 2 | 0

3. Secondary Outcome: TDF and TFV Maximum Concentrations (C-max) in CVF Genital Secretions (ECX and VAG) and TFV Maximum Concentration in Plasma
Description: TDF (tenofovir disoproxil fumarate) and TFV (tenofovir) maximum concentrations (C-max) in CVF (Cervicovaginal Fluid) genital secretions (ectocervix (ECX) and vagina (VAG)) and TFV maximum concentration (C-max) in plasma. PK parameters only measured in TDF IVR subjects, not Placebo IVR subjects.
Time Frame: 1, 3, 7 and 14 days after ring insertion and 2 and 7 days after ring removal
Population: TDF analytical data available for 14 of 15 participants for CVF VAG and CVF ECX. PK parameters only measured in TDF IVR subjects, not Placebo IVR subjects.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | TDF Intravaginal Ring | Placebo Intravaginal Ring
Number analyzed (Participants) | 15 | 0
ng/mL
  C-max CVF VAG TDF: number analyzed (Participants) | 14 | 0
  C-max CVF VAG TDF | 240000 [140000 to 360000] |
  C-max CVF ECX TDF: number analyzed (Participants) | 14 | 0
  C-max CVF ECX TDF | 210000 [81000 to 320000] |
  C-max CVF VAG TFV | 91000 [73000 to 190000] |
  C-max CVF ECX TFV | 85000 [52000 to 170000] |
  C-max Plasma TFV | 1.9 [1.2 to 2.4] |

4. Secondary Outcome: TDF and TFV Time to Maximum Concentrations (T-max) in CVF Genital Secretions (ECX and VAG), and TFV Time to Maximum Concentration in Plasma
Description: TDF (tenofovir disoproxil fumarate) and TFV (tenofovir) time to maximum concentrations (T-max) in CVF (Cervicovaginal Fluid) genital secretions (ectocervix (ECX) and vagina (VAG)), and TFV time to maximum concentration in Plasma. PK parameters only measured in TDF IVR subjects, not Placebo IVR subjects.
Time Frame: 1, 3, 7 and 14 days after ring insertion and 2 and 7 days after ring removal
Population: TDF analytical data available for 14 of 15 participants for CVF VAG and CVF ECX. TFV analytical data available for 12 of 15 participants for Plasma. PK parameters only measured in TDF IVR subjects, not Placebo IVR subjects.
Measure: Median (Inter-Quartile Range); unit: h
Arm/Group | TDF Intravaginal Ring | Placebo Intravaginal Ring
Number analyzed (Participants) | 15 | 0
h
  T-max CVF VAG TDF: number analyzed (Participants) | 14 | 0
  T-max CVF VAG TDF | 6 [3 to 7] |
  T-max CVF ECX TDF: number analyzed (Participants) | 14 | 0
  T-max CVF ECX TDF | 5 [4 to 7] |
  T-max CVF VAG TFV | 14 [1 to 14] |
  T-max CVF ECX TFV | 7 [3 to 14] |
  T-max Plasma TFV: number analyzed (Participants) | 12 | 0
  T-max Plasma TFV | 14 [14 to 14] |

5. Secondary Outcome: TDF AUC0-14 in CVF Genital Secretions (ECX and VAG), TFV AUC0-14 in CVF Genital Secretions (ECX and VAG), and TFV AUC0-14 in Plasma
Description: TDF (tenofovir disoproxil fumarate) AUC0-14 (Area Under the Curve (concentration versus time) days 0-14) in Cervicovaginal Fluid (CVF) genital secretions (ectocervix (ECX) and vagina(VAG)), TFV AUC0-14 in CVF genital secretions (ECX and VAG), and TFV (tenofovir) AUC0-14 in Plasma. PK parameters only measured in TDF IVR subjects, not Placebo IVR subjects.
Time Frame: 1, 3, 7 and 14 days after ring insertion and 2 and 7 days after ring removal
Population: TDF analytical data available for 13 of 15 participants for CVF ECX, and 14 of 15 participants for CVF VAG. TFV analytical data available for 13 of 15 participants for CVF ECX. PK parameters only measured in TDF IVR subjects, not Placebo IVR subjects.
Measure: Median (Inter-Quartile Range); unit: ngxd/mL
Arm/Group | TDF Intravaginal Ring | Placebo Intravaginal Ring
Number analyzed (Participants) | 15 | 0
ngxd/mL
  AUC0-14 (days 0-14), CVF VAG TDF: number analyzed (Participants) | 14 | 0
  AUC0-14 (days 0-14), CVF VAG TDF | 2000000 [690000 to 3200000] |
  AUC0-14 (days 0-14), CVF ECX TDF: number analyzed (Participants) | 13 | 0
  AUC0-14 (days 0-14), CVF ECX TDF | 1300000 [340000 to 2100000] |
  AUC0-14 (days 0-14), CVF VAG TFV | 1100000 [670000 to 2100000] |
  AUC0-14 (days 0-14), CVF ECX TFV: number analyzed (Participants) | 13 | 0
  AUC0-14 (days 0-14), CVF ECX TFV | 970000 [570000 to 1300000] |
  AUC0-14 (days 0-14), Plasma TFV | 9.4 [6.9 to 14.4] |

6. Secondary Outcome: TFV C-ave in Cervical Tissue
Description: TFV (tenofovir) average concentration (C-ave) in cervical tissue. PK parameters only measured in TDF IVR subjects, not Placebo IVR subjects.
Time Frame: before and after 14 days of vaginal ring use
Population: PK parameters only measured in TDF IVR subjects, not Placebo IVR subjects.
Measure: Median (Inter-Quartile Range); unit: ng/mg
Arm/Group | TDF Intravaginal Ring | Placebo Intravaginal Ring
Number analyzed (Participants) | 15 | 0
ng/mg | 5.4 [2.8 to 8.8] |

7. Secondary Outcome: TFV-DP C-ave in Cervical Tissue
Description: TFV-DP (tenofovir diphosphate) average concentration (C-ave) in cervical tissue. PK parameters only measured in TDF IVR subjects, not Placebo IVR subjects.
Time Frame: before and after 14 days of vaginal ring use
Population: PK parameters only measured in TDF IVR subjects, not Placebo IVR subjects.
Measure: Median (Inter-Quartile Range); unit: fmol/mg
Arm/Group | TDF Intravaginal Ring | Placebo Intravaginal Ring
Number analyzed (Participants) | 15 | 0
fmol/mg | 120 [90 to 550] |

ADVERSE EVENTS:
Arm/Group | TDF Intravaginal Ring | Placebo Intravaginal Ring
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 11/15 | 4/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TDF Intravaginal Ring (N=15) | Placebo Intravaginal Ring (N=15)
Vaginal discharge (Reproductive system and breast disorders) | 6 | 1
Intermenstrual bleeding (Reproductive system and breast disorders) | 3 | 3
Pelvic pain (Reproductive system and breast disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes